CLINICAL TRIAL: NCT02801799
Title: Effects of Local Anaesthetic Infusion Rates on Nerve Block Duration. A Randomised, Blinded, Healthy Volunteer Study
Brief Title: Effects of Local Anaesthetic Infusion Rates on Nerve Block Duration
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was comprised of two parts. After the first part we could repudiate our hypothesis. Thus, no reason to carry on with the second part of the trial.
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: FIPRA 1
Record Dates: First submitted 2016-06-03; First posted 2016-06-16 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2016-06

CONDITIONS: Other Acute Postoperative Pain; Pain, Postoperative; Anaesthesia
Keywords: Anaesthesia; Analgesia; Nerve blocks; Peripheral nerve blocks; Regional anaesthesia; therapeutic techniques; ropivacaine; nerve block duration; lower limb; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Infusion group 1 (Active Comparator): Intervention:
  One peri-neural infusion of a fixed volume of ropivacaine 0.2%, administered via a perineurial nerve catheter.
  Infusion rate will be 12 mL/h. This infusion rate is normal clinical practice when administering a perineural infusion of ropivacaine.
  Interventions: Drug: Varying infusion rates of Ropivacaine 0.2%
- Infusion group 2 (Experimental): Intervention:
  One peri-neural infusion of a fixed volume of ropivacaine 0.2%, administered via a perineurial nerve catheter.
  Infusion rate will be 60 mL/h. This infusion rate is experimental.
  Interventions: Drug: Varying infusion rates of Ropivacaine 0.2%
- Infusion group 3 (Experimental): Intervention:
  One peri-neural infusion of a fixed volume of ropivacaine 0.2%, administered via a perineurial nerve catheter.
  Infusion rate will be 300 mL/h. This infusion rate is experimental.
  Interventions: Drug: Varying infusion rates of Ropivacaine 0.2%
- Infusion group 4 (Experimental): Intervention:
  One peri-neural infusion of a fixed volume of ropivacaine 0.2%, administered via a perineurial nerve catheter.
  Infusion rate will be 600 mL/h. This infusion rate is experimental.
  Interventions: Drug: Varying infusion rates of Ropivacaine 0.2%
- Infusion group 5 (Active Comparator): Intervention:
  One peri-neural infusion of a fixed volume of ropivacaine 0.2%, administered via a perineurial nerve catheter.
  Infusion rate will be 1800 mL/h. This infusion rate is normal clinical practice when administering a perineural bolus of ropivacaine.
  Interventions: Drug: Varying infusion rates of Ropivacaine 0.2%

INTERVENTIONS:
Drug: Varying infusion rates of Ropivacaine 0.2% — Participants will receive one nerve catheter adjacent to the common peroneal nerve (trial day 1) and adjacent to the sciatic nerve (trial day 2). Each catheter will be randomly allocated to one of five infusion groups. All peroneal nerve catheters will receive the same volume of ropivacaine 0.2%. All the sciatic nerve catheters will receive the same volume of ropivacaine 0.2%.
  The only inter-group variable will be the infusion rate. The fixed volume of ropivacaine will be determined in a separate study ('The Volume Study'), which is also part of the project: 'A novel technique for reliable, precise and safe postoperative management'.
  The largest volumes tested in "The Volume Study" are 30 mL for the sciatic nerve and 20 mL for the common peroneal nerve. Therefore the highest volume for the two intervention days cannot exceed 30 mL (150 mg of ropivacaine).
  We will ensure constant infusion rate and precise delivery of LA by using an electronic infusion pump and a nerve catheter.

SUMMARY:
This trial is a part of the project: 'A novel technique for reliable, precise and safe postoperative pain management' (project no. 65-2014-3).

The purpose of the trial is to investigate the effects of changing peri-neural infusion rates of ropivacaine 0.2% on the duration of nerve block.

Intervention:

Two intervention-days. Each day a peri-neural infusion of a fixed volume of ropivacaine 0.2% is to be infused in one of five infusion rates, using a peri-neural catheter.

Intervention day 1: Focus on the common peroneal nerve. Intervention day 2: Focus on the sciatic nerve.

DETAILED DESCRIPTION:
This trial is a part of the project: 'A novel technique for reliable, precise and safe postoperative pain management' (project no. 65-2014-3). Results will contribute to the development of an electrical disposable infusion pump manufactured by Ferrosan Medical Devices (FEMD). It is made up of two half's; first intervening day focuses on the common peroneal nerve, second intervening day focuses on the sciatic nerve.

Hypothesis:

The infusion rate of a single peri-neural injection of LA does not influence the duration of lower limb nerve blocks.

Trial objective:

We wish to compare five peri-neural infusion rates of LA as an independent factor of the duration of the nerve block, in the sciatic nerve and the common peroneal nerve, in healthy volunteers.

The slowest infusion will simulate a standard infusion rate for continuous infusion. The fastest infusion will simulate a standard bolus rate when administering a LA bolus. The three infusions in between are to our knowledge new alternative infusion rates.

Trial design:

Prospective, randomised, blinded, single centre, healthy volunteer study.

Intervention medication:

Ropivacaine 0.2%

Detailed description of the intervention:

Baseline measurements and safety precautions The volunteers will meet at the Clinical Research Unit, Nordsjællands Hospital Hillerød, following a six-hour fast. After baseline measurements, we will insert a peripheral intravenous catheter and start continuous pulse oximetry.

Placing the catheters

We will insert one peri-neural catheter at each of the intervention days:

1. Adjacent to common peroneal nerve on the non-dominant side. The participant will be supine on the dominant side.
2. Adjacent to the proximal part of the sciatic nerve on the non-dominant side. The participant will be in prone position.

An expert in peripheral nerve blocks will perform catheter placement in a sterile manner, using an ultrasound (US) guided short-axis, needle in-plane technique and a high frequency linear transducer.

Using lidocaine 1% we will raise a small skin wheal at the needle entry point and anaesthetise the trajectory of the catheter needle.

3 mL of isotonic saline will be deposited in the peri-neural tissue before placing the catheter. This ensures optimal conditions for placing the nerve catheters.

Successful catheter orifice placement will be ensured by visually confirmation of the echogenic markings of the catheter and a 2 mL isotonic saline injection through the orifice.

After insertion, a sterile dressing will be placed, covering the catheters. Absorption from the peri-neural space We will verify full absorption of the isotonic saline in the peri-neural space by US. When full absorption is confirmed, members of the investigator team must leave the room.

Preparation for infusion A trial-affiliated nurse that is not part of the investigator team will prepare one 50 ml syringe, imbibing 30 mL of ropivacaine 0.5%. This step will be over-looked by a random, un-affiliated college to ensure double-control of correct intervention.

Peri-neural infusions

The trial-affiliated nurse will connect a transfusion hose and mount the syringe in the infusion pump. The nurse will activate a 2 mL bolus on the infusion pump, flushing the transfusion hose and then connect the transfusion hose to the nerve catheter. The trial-affiliated nurse will open the opaque envelope that matches the participant and prepare the infusion and administration as prescribed according to one of the five infusion groups:

Infusion Groups and Infusion rates [mL/hour] / [mL/min] IG1 12 / 0.2 IG2 60 / 1 IG3 300 / 5 IG4 600 / 10 IG5 1800 / 30

This step will be over-looked by a random, un-affiliated college to ensure double-control of correct intervention.

The trial-affiliated nurse will start the infusion and the investigator team is allowed back in.

Measuring outcomes

The outcomes will be measured in the following way:

1. Measuring length of neural exposure to ropivacaine five times, according to calculated infusion time.
2. Finding sensory onset time by five minutes intervals.
3. Grading the degree of sensory nerve block after registered onset time.
4. Grading the degree of motor nerve block after the catheter has been removed. Investigators will start testing for sensory onset time 10 minutes after start of infusion.

All outcomes and outcome measurements are described in detail in the section "Outcomes".

To ensure that manipulation of the catheter will not affect the distribution and absorption of LA, the catheters will not be removed until 30 minutes after end of the slowest infusion.

We estimate the mean and maximal duration of the sciatic nerve block to be seventeen and twenty-four hours, respectively15,20-24. Consequently, the duration of each study day is expected to be no more than twenty-four hours. The volunteer will be offered discharge at the time of complete nerve block remission. In exceptional cases of incomplete nerve block remission within twenty-four hours, the volunteer will be asked to stay admitted for continued testing.

At all times, adequately trained health-care personnel with rescue medicine and resuscitation equipment at hand will be in proximity to the volunteer.

Intervention related information

* Members of the investigator team who are medical doctors and skilled in performing US-guided peripheral nerve blocks will insert the peripheral nerve catheters.
* The Certa Catheter™ will be used as recommended by the manufacturer.
* Study medications as well as medications used for concomitant care will be handled according to local guidelines and provided and stored by The Department of Anaesthesiology and Intensive Care, Nordsjællands Hospital Hillerød via the hospital pharmacy until its use. During the study period, once a week, medications will be taken from the locked storage of the Post Anaesthesia Care Unit to the locked storage of the Clinical Research Unit, Nordsjællands Hospital Hillerød.
* All personnel involved in conduction of the intervention is adequately educated and experienced in performing basal resuscitation.

Discontinuance

The intervention will be discontinued if:

* the participant withdraws consent.
* the participant experiences symptoms of LA systemic toxicity.
* the participant exhibits symptoms of an allergic reaction.
* there is any suspicion of nerve injury In addition to these specific reasons, adverse reactions of any severity and lack of compliance to instructions may cause discontinuance.

Concomitant care

1. Sedation If indicated, investigators will administer midazolam (0.03 mg/kg).
2. Treatment of pain Skin infiltration anaesthesia will be necessary when inserting the catheters the investigator will administer a maximum of 2 mL of lidocaine 1 mg/mL as a subcutaneous papilla, ensuring non-influential proximity to the sciatic nerve. If the participant experiences unbearable pain during insertion of the catheters administration of a standard short acting, intravenous analgesic (0.5-1.5 mg of Rapifen depending on weight, age and administration and sedation) will be allowed.
3. General care During the trial day the participant will receive meals, snacks and tap water. The participant will have a bed available at all times, placed in a two-person room.

Sample size:

To be able to detect a difference with a power of 80% and a margin of error of 5%, when testing our null-hypothesis, we need the participant number in each infusion group to be larger than 10.9. Thus, each infusion group will have at least 11 participants, making the sample size for each intervention-day at least 55 and the total sample size at least 110. To account for potential dropouts, we wish to include 60 healthy volunteers for each intervention-day, totalling 120 healthy volunteers.

Sequence generation:

all study numbers will be block-randomised electronically by a non-trial-affiliated person to one of the five equally sized infusion groups of the first intervention day. This step will be repeated before the second intervention day.

Allocation concealment mechanism:

Until study termination of FIPRA 1, allocation sequence will be concealed to the investigator team and noted electronically on a computer belonging to the Research Unit, Department of Anaesthesiology and Intensive Care, Nordsjællands Hospital Hillerød.

Blinding:

All volunteers and outcome assessors will be blinded to the LA administration and infusion procedures.

Harms Unanticipated problems involving risks to subjects or others, adverse events and adverse reactions will be reviewed and reported in accordance to the current thinking by The Danish Unit for Good Clinical Practice and The Danish Medicines Agency. The reporting will happen within the timeframe stated by the order of clinical trials with drugs on human subjects (order #295 of 26th of April 2004 in The Danish Law)

Research ethics approval This trial will be conducted according to guidelines provided by The International Council for Harmonisation (ICH), The Danish Unit for Good Clinical Practice (GCP) and The Declaration of Helsinki3. We will register/announce the study at The Scientific Ethics Committee, The Danish Health and Medicines Authority, The Danish Data Protection Agency, The Danish Unit for Good Clinical Practice and at clinicaltrials.gov. The trial is initiated after all official approvals have been given.

Access to data During the trial only the investigators will have access to CRFs and the raw data material. After the trial the primary investigator, sponsor and supervisor will have access to the full trial dataset.

The data will be stored for 5 years by The Research Unit, Department of Anaesthesiology and Intensive Care, Nordsjællands Hospital Hillerød.

As part of the Co-funding agreement between Innovation Fund Denmark, NOH and FEMD (Journal no. 65-2014-3), results from this study will contribute to the development of an electronic disposable infusion pump manufactured by FEMD. Furthermore, before publishing, FEMD, has the right to review the manuscript to ensure that no intellectual properties (IP's) belonging to FEMD are published. If so, FEMD may claim additional thirty days before submission to apply for new patent or other protection of IP. FEMD is not allowed to comment or change any other parts of the manuscript.

The Research Unit, Department of Anaesthesiology and Intensive Care, NOH retains ownership of all raw clinical data and may use data as they see fit.

ELIGIBILITY:
Inclusion criteria

1. Male or female ≥18, ≤ 64 years of age
2. ASA classification17 ≤ II

Exclusion criteria

1. BMI ≤ 18 or ≥ 30 kg/m2
2. Body weight ≤ 37.5 kg
3. Former surgery to the lower extremities
4. Peripheral nerve disease, including polyneuropathy and diabetes
5. Allergy to local anaesthetics
6. Pregnancy or breastfeeding
7. Enrolment in other investigational drug studies or recent clinical trials that may interfere with this study
8. Habitual use of any kind of analgesic treatment
9. Anatomic abnormalities preventing successful US-guided Certa Catheter™ insertion.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2016-11-23 (Actual); Study Completion 2016-12-09 (Actual)

PRIMARY OUTCOMES:
Duration of insensitivity towards cold | Until nerve block remission (expected to be less than 24 hours).
  Measuring insensitivity towards cold using cutaneous application of a round, cooled glass container, stored in a refrigerator (5°C). The time of normal sensation is subtracted the time of onset.
  This non-invasive measurement is a well-established way to evaluate the presumed anaesthetic effect of LA. It will be performed in the cutaneous innervation of the common peroneal nerve and the sciatic nerve accordingly. It will be measured in hours.

SECONDARY OUTCOMES:
Length of neural exposure to ropivacaine | During drug administration, no longer than 150 minutes.
  Spread of ropivacaine along the common peroneal nerve and the sciatic nerve will be measured five times during the infusion of ropivacaine, using US. According to the volume to be infused, each of the five infusion groups will have a designated infusion-time. For each infusion, we will perform this measurement at each of these five calculated time points. Like this every participant will have a US scan five times.
Time to onset of sensory nerve block | From start of infusion until onset of sensory nerve block or for no more than three hours
  Time from start of infusion until first positive test, measured in minutes.
Degree of motor nerve block | Until nerve block remission (expected to be less than 24 hours).
  In an upright position and with a sturdy county as support, the degree of motor nerve block will be measured using a normal everyday activation of the lower leg; A toe and a heel raise, testing the common peroneal nerve via activation of the anterior tibial muscle and the tibial nerve via activation of the gastrocnemius muscle, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel H. Madsen, MD, Principal Investigator — Research Unit, Department of Anaesthesiology and Intensive Care, Nordsjaellands Hospital Hilleroed
Locations (1):
- Research Unit, Department of Anaesthesiology and Intensive Care, Nordsjaellands Hospital Hilleroed, Hilleroed, Capital Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
No matter the outcome of this trial tre results will be available at ClinicalTrials.gov, EudraCT.ema.europa.eu and will as far as possible, be published in a scientific paper of relevance for regional anesthesia.

REFERENCES:
- [Derived] Madsen MH, Christiansen CB, Rothe C, Andreasen AM, Lundstrom LH, Lange KHW. Local Anesthetic Injection Speed and Common Peroneal Nerve Block Duration: A Randomized Controlled Trial in Healthy Volunteers. Reg Anesth Pain Med. 2018 Jul;43(5):467-473. doi: 10.1097/AAP.0000000000000759. PMID 29570501